CLINICAL TRIAL: NCT00272649
Title: A Phase I/II Study Testing the Biologic Activity and Safety of AGS-003 as an Immunotherapeutic in Subjects With Newly Diagnosed Stage IV Renal Cell Carcinoma
Brief Title: Study Testing the Biologic Activity and Safety of an Immunotherapeutic in Patients With Newly Diagnosed Stage IV Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Argos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGS-003-004; Bukowski-8077; Logan-0506-05; Drabkin-05-0167; White-04-05-01A; Figlin-05-03-099-01; NCT00309829 (obsolete NCT alias)
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Renal Cell Carcinoma
Keywords: Kidney cancer; Renal cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Single Arm study
  Interventions: Biological: AGS-003

INTERVENTIONS:
Biological: AGS-003 — Dendritic cell, autologous cellular immunotherapy. (Arcelis platform)
  Other Names: Dendritic Cell Immunotherapeutic

SUMMARY:
The purpose of this trial is to examine the safety, feasibility, immunological response, and clinical antitumor activity of multiple administrations of dendritic cell Immunotherapeutic to patients with newly diagnosed with metastatic kidney cancer

DETAILED DESCRIPTION:
In this study, a new Immunotherapeutic production process will be used that shows evidence of potentially much higher biologic activity in pre-clinical studies than the production process used in a previous study (clinical protocol MB-002-003). While both processes are based on individual subject autologous tumor RNA and autologous monocyte derived DCs, the maturation of DCs in this newly modified process involves an altered regimen of culture with cytokines. In addition, huCD40L mRNA is added to the autologous expanded tumor total mRNA for electroporation. These changes promise a much improved migration, and activity profile of the DC-Immunotherapeutic product in RCC subjects.

ELIGIBILITY:
Inclusion Criteria:

* Have a new diagnosis of metastatic renal cell carcinoma;
* Measurable disease
* Must be at least 18 years or older;
* Have a scheduled unilateral nephrectomy or excisional biopsy/metastasectomy
* ECOG of 0 or 1;
* Free of brain metastases by CT or MRI;
* Normal renal function in contralateral kidney;
* Male or non-pregnant/non-lactating female on appropriate birth control methods while on study;
* Clinically acceptable screening results.
* No immunosuppressive therapy not limited to corticosteroids (including topical steroids or steroid containing inhalers), azathioprine cyclosporine two months prior to study entry;
* No active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
1. Measure tumor response by RECIST as CR, PR, SD, PD. 2. Measure T-cell responses to vaccination using induction vaccination regimens. | 24 weeks

SECONDARY OUTCOMES:
Assess safety of multiple administrations of the Immunotherapeutic in subjects with newly diagnosed, metastatic Renal Cell Cancer Assess Overall Survival and Time to progression | 24 weeks plus follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Terry Chew, MD, Study Chair — Argos Therapeutics
Locations (10):
- United States (8):
  - UCLA Kidney Cancer Program, Los Angeles, California
  - Univ. of Colorado Health Science Center - Division of Medical Oncology, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - The Indiana University Cancer Center/IUPUI, Indianapolis, Indiana
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Carolinas Medical Center/Blumenthal Cancer Center, Charlotte, North Carolina
  - Earle A. Chiles Research Institute, Portland, Oregon
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- See also: Kidney Cancer Association — http://www.nkca.org